CLINICAL TRIAL: NCT03986190
Title: Family-based eHealth Obesity Prevention Intervention for Hispanic Adolescents
Brief Title: Healthy Juntos Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sara StGeorge, Assistant Professor of Public Health Sciences, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20160415; K01HL133521 (NIH)
Record Dates: First submitted 2019-06-11; First posted 2019-06-14 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Obesity; Activity, Motor; Diet, Healthy; Sedentary Behavior
Keywords: Hispanic; family; digital health; obesity prevention; physical activity; nutrition
MeSH Terms: conditions — Obesity; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Juntos Intervention Condition (Experimental): Parent-adolescent dyads randomized to the Healthy Juntos intervention condition will access a program that includes didactic, behavioral, and positive parenting content from their smartphones for 8 weeks.
  Interventions: Behavioral: Healthy Juntos
- Control Group (No Intervention): This group will receive a digital standard of care - a list of publicly available lifestyle apps and websites which they may access at their discretion.

INTERVENTIONS:
Behavioral: Healthy Juntos — Parent-adolescent dyads will log in to a secured website for a total of eight weeks. The intervention will be delivered primarily through smartphones and will include didactic content on healthy lifestyle behaviors (for parents/adolescents), family behavior change content for setting weekly goals and self-monitoring health behaviors (for parents/adolescents), and positive parenting content (for parents only), all of which were developed in accordance with participant feedback based on formative intervention development work. In addition, and to increase participant compliance/reduce attrition often observed in digital health interventions, human support ("supportive accountability") will be provided. Specifically, each family will be assigned a "coach" who will use video conferencing software to engage in weekly 15-30 minute sessions regarding the family's progress throughout the intervention period.
  Arms: Healthy Juntos Intervention Condition

SUMMARY:
The purpose of the study is to assess the feasibility, acceptability, and preliminary effects of a digital (web and mobile phone-based) program to improve physical activity levels and quality dietary intake among Hispanic parent-adolescent dyads.

ELIGIBILITY:
Inclusion criteria:

1. Female and male adolescents whose primary caregiver self-identifies as Hispanic
2. Adolescent is between the ages of 12-15;
3. Adolescent lives with an adult primary caregiver willing to participate;
4. Both parent and adolescent have smartphone/mobile device with internet access;
5. Adolescent does not meet recommendations for fruit and vegetable intake (proxy for overall diet quality) as determined by a validated two-item screener;
6. Adolescent does not meet physical activity guidelines as determined by responses on a validated two-item screener AND self-reports engaging in >2 hours/day of screen time (proxy for overall sedentary behavior) using three items.

Exclusion Criteria:

1. Adolescent's body mass index for age and gender is ≥ 95th percentile ("obese" range);
2. Adolescent has a chronic medical condition (e.g., type 2 diabetes) that requires intensive lifestyle modification;
3. Adolescent has a diagnosed developmental delay that would interfere with understanding program materials;
4. Parent or adolescent has a diagnosed medical or psychiatric condition and is currently taking medications that would interfere with changes to physical activity or diet (e.g., adolescent is diagnosed with Attention Deficit Hyperactivity Disorder and is currently on stimulant medication);
5. Family is planning to move out of the South Florida during the study follow-up period

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara M St George, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 50 parent-adolescent dyads were enrolled and randomized.
Period: Overall Study
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Started | 50 | 50
Adolescents Started | 25 | 25
Parents Started | 25 | 25
Adolescents Completed | 19 | 25
Parents Completed | 19 | 25
Completed | 38 | 50
Not Completed | 12 | 0
Not completed — Withdrawal by Subject | 12 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Juntos Intervention Condition | Control Group | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Customized [Mean (Standard Deviation); unit: years] — Population: A total of 50 participants were included in each arm. Given the nature of the intervention being dyadic we have included 25 parents and 25 adolescents for each group to provide each group's age.
  years
    Adolescents: number analyzed (Participants) | 25 | 25 | 50
    Adolescents | 13.70 (1.02) | 14 (1.21) | 13.80 (1.11)
    Parents: number analyzed (Participants) | 25 | 25 | 50
    Parents | 41.90 (7.54) | 43.90 (6.25) | 42.90 (6.92)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: A total of 50 participants were included in each arm. Because the study enrolled dyads, comprised of one parent and one adolescent, we enrolled 25 parents and 25 adolescents into each group and summarized sex/gender separately for parents and adolescents.
  Participants
    Adolescents: number analyzed (Participants) | 25 | 25 | 50
    Adolescents: Male | 13 | 12 | 25
    Adolescents: Female | 12 | 13 | 25
    Parents: number analyzed (Participants) | 25 | 25 | 50
    Parents: Male | 2 | 4 | 6
    Parents: Female | 23 | 21 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 50 | 50 | 100
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Physical Activity [Mean (Standard Deviation); unit: Minutes/day] — Population: Results are displayed separately for parents and adolescents.
  Minutes/day
    Adolescents MVPA out-of school: number analyzed (Participants) | 25 | 25 | 50
    Adolescents MVPA out-of school | 13.20 (1.94) | 12.72 (1.84) | 12.96 (1.88)
    Adolescents MVPA at school: number analyzed (Participants) | 25 | 25 | 50
    Adolescents MVPA at school | 12.13 (1.50) | 12.35 (1.86) | 12.24 (1.68)
    Adolescents MVPA during the weekend: number analyzed (Participants) | 25 | 25 | 50
    Adolescents MVPA during the weekend | 10.89 (1.31) | 11.17 (1.53) | 11.03 (1.42)
    Parents MVPA: number analyzed (Participants) | 25 | 25 | 50
    Parents MVPA | 56.88 (64.70) | 57.83 (59.56) | 57.34 (61.56)
Fruit and Vegetable Intake [Mean (Standard Deviation); unit: cups/day] — Population: Results are displayed by separately for parents and adolescents.
  cups/day
    Adolescents vegetables intake including legumes and no fries: number analyzed (Participants) | 25 | 25 | 50
    Adolescents vegetables intake including legumes and no fries | 1.11 (0.43) | 1.10 (0.4) | 1.10 (0.41)
    Adolescents fruit intake: number analyzed (Participants) | 25 | 25 | 50
    Adolescents fruit intake | 0.85 (0.76) | 0.93 (0.69) | 0.89 (0.72)
    Parents vegetables intake including legumes and no fries: number analyzed (Participants) | 25 | 25 | 50
    Parents vegetables intake including legumes and no fries | 1.32 (0.38) | 1.33 (0.46) | 1.33 (0.42)
    Parents fruit intake: number analyzed (Participants) | 25 | 25 | 50
    Parents fruit intake | 0.75 (0.28) | 0.77 (0.30) | 0.76 (0.29)
Adolescents Sedentary Behavior Out-of-school [Mean (Standard Deviation); unit: Minutes/day] — Population: Results are displayed separately for parents and adolescents.
  Minutes/day
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 58.73 (2.20) | 58.11 (2.82) | 58.42 (2.52)
Parents Sedentary Behavior [Mean (Standard Deviation); unit: Sitting hours/day] — Population: Results are displayed separately for parents and adolescents
  Sitting hours/day
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 4.28 (2.95) | 3.26 (2.37) | 3.78 (2.70)

OUTCOME MEASURES:

1. Primary Outcome: Change in Adolescents Physical Activity
Description: Adolescents will self-report physical activity using the Youth Activity Profile.
Time Frame: Baseline, up to 2 months
Population: Analyzed number corresponds to those that completed measurements. Number is lower due to drop-off of participants.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Number analyzed (Participants) | 19 | 25
minutes/day
  MVPA out-of school: number analyzed (Participants) | 13 | 24
  MVPA out-of school | 0.62 (1.31) | -0.13 (1.49)
  MVPA at school: number analyzed (Participants) | 13 | 23
  MVPA at school | -0.18 (1.96) | -0.05 (1.06)
  MVPA during the weekend: number analyzed (Participants) | 18 | 24
  MVPA during the weekend | 5.29 (8.04) | -2.40 (15.77)

2. Primary Outcome: Change in Adolescent Sedentary Behavior
Description: Adolescents will self-report sedentary behavior using the Youth Activity Profile.
Time Frame: Baseline, 2 months
Population: Analyzed number corresponds to those that completed measurements. Number is lower due to drop-off.
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Number analyzed (Participants) | 19 | 25
minutes/day | -0.35 (11.25) | -3.08 (13.61)

3. Primary Outcome: Change in Adolescents Dietary Intake (i.e., Fruits/Vegetables)
Description: Adolescents will self-report dietary intake using the NHANES Dietary Screener Questionnaire. Cup equivalents of fruits and vegetables will be calculated using a scoring algorithm developed by the National Cancer Institute.
Time Frame: Baseline, 2 months
Population: Analyzed number corresponds to those that completed measurements. Number is lower due to drop-off from baseline to T2 assessment.
Measure: Mean (Standard Deviation); unit: cups/day
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Number analyzed (Participants) | 19 | 25
cups/day
  Vegetables intake including legumes and no fries: number analyzed (Participants) | 18 | 22
  Vegetables intake including legumes and no fries | 0.33 (0.99) | -0.17 (0.85)
  Fruit intake: number analyzed (Participants) | 19 | 24
  Fruit intake | 0.13 (1.06) | -0.16 (0.73)

4. Primary Outcome: Change in Adolescents Dietary Intake (Sugar)
Description: Adolescent-parent dyads will self-report dietary intake using the NHANES Dietary Screener Questionnaire. Teaspoon equivalents of added sugars.
Time Frame: Baseline, up to 2 months
Population: Difference at control group is due to lost of follow-up.
Measure: Mean (Standard Deviation); unit: Teaspoon per day
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Number analyzed (Participants) | 19 | 25
Teaspoon per day | 1.91 (9.46) | 1.53 (7.50)

5. Secondary Outcome: Change in Parent Physical Activity.
Description: Parents will self-report physical activity using the International Physical Activity Questionnaire.
Time Frame: Baseline, up to 2 months
Measure: Mean (Standard Deviation); unit: minutes/day
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Number analyzed (Participants) | 18 | 23
minutes/day | 38.82 (60.01) | 38.26 (75.49)

6. Secondary Outcome: Change Parent Sedentary Behavior
Description: Parents will self-report their sitting time using a single item from the International Physical Activity Questionnaire
Time Frame: Baseline, up to 2 months
Measure: Mean (Standard Deviation); unit: sitting hours/day
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Number analyzed (Participants) | 18 | 23
sitting hours/day | -0.04 (1.92) | 0.34 (2.45)

7. Secondary Outcome: Change in Parents Dietary Intake (i.e., Fruits/Vegetables)
Description: Parents will self-report dietary intake using the NHANES Dietary Screener Questionnaire. Cup equivalents of fruits and vegetables will be calculated using a scoring algorithm developed by the National Cancer Institute.
Time Frame: Baseline, up to 2 months
Population: Difference is total numbers due to drop-off.
Measure: Mean (Standard Deviation); unit: cups/day
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Number analyzed (Participants) | 19 | 25
cups/day
  Vegetables intake including legumes and no fries: number analyzed (Participants) | 18 | 24
  Vegetables intake including legumes and no fries | 0.21 (0.33) | -0.02 (0.46)
  Fruit intake | 0.06 (0.26) | -0.01 (0.38)

8. Secondary Outcome: Change in Parents Dietary Intake (Sugar)
Description: Parents will self-report dietary intake using the NHANES Dietary Screener Questionnaire. Teaspoon equivalents of added sugars.
Time Frame: Baseline, up to 2 months
Measure: Mean (Standard Deviation); unit: teaspoon/day
Arm/Group | Healthy Juntos Intervention Condition | Control Group
Number analyzed (Participants) | 19 | 23
teaspoon/day | -1.25 (2.93) | 1.28 (5.53)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Healthy Juntos Intervention Condition | Control Group
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/90/NCT03986190/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03986190/ICF_001.pdf